CLINICAL TRIAL: NCT05586568
Title: A Drug-drug Interaction Study Evaluating the Pharmacokinetic Effects of Itraconazole or Rifampin or Esomeprazole on XZP-3621 Tablets in Healthy Subjects
Brief Title: Drug-drug Interaction Study of XZP-3621 Tablet
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XZP-3621-1003
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-08

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Rifampin; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- XZP-3621 tablet and itraconazole oral liquid (Experimental)
  Interventions: Drug: XZP-3621 tablet and itraconazole oral liquid (for Arm1)
- XZP-3621 tablet and Rifampicin capsules (Experimental)
  Interventions: Drug: XZP-3621 tablet and Rifampicin capsules (For Arm 2)
- XZP-3621 tablet and esomeprazole tablet (Experimental)
  Interventions: Drug: XZP-3621 tablet and esomeprazole tablet (For Arm3)

INTERVENTIONS:
Drug: XZP-3621 tablet and itraconazole oral liquid (for Arm1) — There are 2 periods, for the 1st period, the subjects will only take XZP-3621 tablets QD on Day1. For period 2,the subjects will take itraconazole from Day11 to Day13，they will take itraconazole in combinaiton with XZP-3621 on Day14，then take itraconazole only, from Day15 to Day27.
  Arms: XZP-3621 tablet and itraconazole oral liquid
Drug: XZP-3621 tablet and Rifampicin capsules (For Arm 2) — There are 2 periods, for the 1st period, the subjects will only take XZP-3621 tablets qd on Day1 . For period 2,the subjects will take Rifampicin from Day11 to Day17，they will take Rifampicin in combinaiton with XZP-3621 on day18，then take Rifampicin only, from Day19 to Day26.
  Arms: XZP-3621 tablet and Rifampicin capsules
Drug: XZP-3621 tablet and esomeprazole tablet (For Arm3) — There are 2 periods, for the 1st period, the subjects will only take XZP-3621 tablets QD on Day1 . For period 2,the subjects will take esomeprazole from Day11 to Day 15，they will take esomeprazole in combinaiton with XZP-3621 on Day16.
  Arms: XZP-3621 tablet and esomeprazole tablet

SUMMARY:
This is an open-label, single center, 2 period, one sequence study to investigate the potential drug drug interaction between itraconazole or rifampin or esomeprazole and XZP-3621 tablet.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18-65 years (including boundary values);
2. Male weight ≥50kg, female weight ≥45kg, body mass index (bmi) in the range of 19-28 kg/m2 (including boundary value);
3. No mental abnormalities, cardiovascular system, nervous system, respiratory system, digestive system, urinary system, History of systemic, endocrine and metabolic abnormalities;
4. The subject and his/her partner agreed to use effective contraception and had no plans to donate sperm or eggs from the time of trial screening until 6 months after the last dose. Women of childbearing age must have a negative blood pregnancy test before the first dose;
5. The subjects should be able to communicate well with the researchers, understand and comply with the requirements of the study, and understand and sign the informed consent.

Exclusion Criteria:

* 1. Allergy (allergy to two or more substances) or known allergy to XZP-3621 or similar drugs (Group 1 (itraconazole group) excluded patients with history of allergy to itraconazole or similar drugs; group 2 (rifampicin group) excluded patients with allergy to rifampicin or its similar antibacterial drugs); The third group (esomeprazole group) excluded patients with esomeprazole or similar drug allergy history];

  2.During screening, there are clinical significant abnormal results in Physical examination, laboratory tests, 12-lead electrocardiogram, Anteroposterior and lateral chest x-ray examination or abdomen B ultrasound examination (including thyroid dysfunction with clinical significance)

  3. Frequent use of sedation, sleeping pills or other addictive drugs within 6 months before enrollment;

  4. Patients with a history of drug abuse or positive urine drug screening within 12 months before enrollment;

  5. Smokers who smoked more than 5 cigarettes per day in the 3 months before screening, or who could not stop using any tobacco products during the study;

  6. Alcohol breath test positive o regular drinkers within 6 months before enrollment, drinking more than 3 units per day, or more than 21 units of alcohol per week(1 unit is equivalent to a 350-ml bottle beer or 120 mL liquor or 30 mL spirits (above 50°)];

  7. Use any prescription drugs or traditional Chinese medicine within 4 weeks before enrollment, and/or use any OTC drugs or food supplements (including vitamins, calcium tablets, etc.) within 2 weeks before the first dose;

  8. Participated in other clinical trials and used investigational drugs within 3 months before enrollment;

  9. Those who received live vaccine within 2 weeks before the first dose, or planned to receive live vaccine during the study or within 7 days after the study was completed;

  10. Blood donation or blood loss of 400 mL within 3 months before enrollment, or blood transfusion; Blood donation (including component blood donation) or blood loss of 200 mL within 1 month before enrollment;

  11. Have a history of major disease or major surgery or trauma within 3 months before screening;

  12. Gastrointestinal disease causing clinically significant symptoms such as nausea, vomiting, diarrhea, or malabsorption syndrome, or a history of severe vomiting or diarrhea within one week before enrollment;

  13. Female subjects during pregnancy and lactation and female subjects of reproductive age who cannot take contraception as required;

  14. HBsAg, HCV Ab, Treponema pallidum antibody, HIV Ab test results are positive;

  15. Those who have special dietary requirements (including lactose intolerance) and are unable to comply with the provided diet and corresponding regulations;

  16. Subjects refused to discontinue any beverage or food containing xanthine derivatives, such as caffeine (coffee, tea, cola, chocolate, etc.) for 48 hours before the first dose and until the end of the study;

  17. Use of any drug that inhibits or induces hepatic metabolism (inducer) within 30 days prior to the first dose such as: barbiturates, carbamazepine, phenytoin sodium, rifamequine; Inhibitors such as cimetidine, Cyclosporine, macrolides, verapamil, quinolones, pyrroles, etc.);

  18. Use of proton pump inhibitor (PPI) drugs within 7 days before the first dose(eg: Rabeprazole, pantoprazole, esomeprazole, etc.).

  19. Ingested or planned ingestion of grapefruit or grapefruit-related citrus within 14 days before the first dose Fruit (such as lime, grapefruit), star fruit, papaya, pomegranate or above fruit products;

  20. Those who cannot tolerate blood collection by venipuncture or whose blood vessels are in poor condition;

  21. Other subjects deemed unsuitable to participate in the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-08-02 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration versus time curve of XZP-3621 and its metabolite in plasma (AUC) (Part 1a and Part1b) | Up to nearly 1 month.
  To determine the AUC of XZP-3621 and its metabolite.
Maximum serum concentration (Cmax) of XZP-3621 and its metabolite. | Up to nearly 1 week.
  To determine the maximum serum concentration (Cmax) of XZP-3621 and its metabolite.

SECONDARY OUTCOMES:
Time of Maximum observed serum concentration (Tmax) of XZP-3621 and its metabolite . | Up to nearly 1 week.
  To determine the Tmax of XZP-3621 and its metabolite.
Serum Half-life (T-HALF) of XZP-3621 and its metabolite . | Up to nearly 1 week.
  To determine the t1/2 of XZP-3621 and its metabolite .
Number of patients with adverse events and serious adverse events. | Up to nearly 2 months.
  Number of patients who experienced an adverse event or serious adverse events.
Severity of adverse events and serious adverse events. | Up to nearly 2 months.
  Severity of the adverse events or serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China